CLINICAL TRIAL: NCT06942858
Title: Mechanisms of Deep Transcranial Magnetic Stimulation Enhances the Efficacy of Cognitive-behavioral Therapy (CBT) by Modulating Anterior Cingulate Cortex in Patients With Anorexia Nervosa
Brief Title: Mechanisms of Deep Transcranial Magnetic Stimulation in Enhancing Cognitive-Behavioral Therapy for Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Jue CHEN, Director of Psychosomatic Department in Shanghai Mental Health Center, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82471573
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Feeding and Eating Disorders
Keywords: anorexia nervosa; Deep transcranial magnetic stimulation; anterior cingulate cortex
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT+dTMS treatment group (Experimental): CBT+dTMS treatment group has 55 patients. Each patient receives 12 individual sessions of CBT for 50 minutes 2 times per week for 6 weeks. dTMS intervention use real coils, targeting ACC, given 5 times per week (Monday to Friday) for 6 consecutive weeks.
  Interventions: Device: Deep transcranial magnetic stimulation; Behavioral: cognitive behavior therapy; Other: Basic treatment
- CBT+pseudo-stimulation group (Active Comparator): CBT+Pseudo-stimulation group has 55 patients. Each patient receives 12 individual sessions of CBT for 50 minutes 2 times per week for 6 weeks. dTMS intervention uses sham coils (with the same parameters as real dTMS and generating the same noise as real coils, but without the magnetic field). It is given 5 times per week (Monday to Friday) for 6 consecutive weeks.
  Interventions: Behavioral: cognitive behavior therapy; Device: Sham deep transcranial magnetic stimulation; Other: Basic treatment

INTERVENTIONS:
Device: Deep transcranial magnetic stimulation — M-100 Ultimate pulsed magnetic field stimulator is used for dTMS treatment. The coil is positioned 4 cm anterior to the scalp point and the foot motor cortex, corresponding to the ACC. A naturally cold HF001A coil is used to obtain a greater depth of stimulation, up to about 6 cm subcortical. The coil is an integrated coil for true and false stimulation loops. The intervention protocol is as follows: 30 treatments are given 5 times per week (Monday to Friday) for 6 consecutive weeks. Intervention mode: stimulation frequency 20Hz, stimulation intensity 100% RMT, number of serial pulses 50, sequence interval 20s, a total of 40 trials, 2000 pulses, stimulating the left and right ACC respectively.
  Arms: CBT+dTMS treatment group
Behavioral: cognitive behavior therapy — Each patient receives 12 individual sessions of 50 minutes twice a week for 6 weeks.The CBT therapists are nationally registered psychotherapists with systematic professional training and uniform training in CBT for anorexia nervosa to ensure consistency. They are also supervised by a CBT supervisor at the end of each session.
Device: Sham deep transcranial magnetic stimulation — M-100 Ultimate pulsed magnetic field stimulator is used for dTMS treatment. The coil is positioned 4 cm anterior to the scalp point and the foot motor cortex, corresponding to the ACC (The sham coil has the same parameters as real dTMS and generating the same noise as real coils, but without the magnetic field). A naturally cold HF001A coil is used to obtain a greater depth of stimulation, up to about 6 cm subcortical. The intervention protocol is as follows: 30 treatments are given 5 times per week (Monday to Friday) for 6 consecutive weeks. Intervention mode: stimulation frequency 20Hz, stimulation intensity 100% RMT, number of serial pulses 50, sequence interval 20s, a total of 40 trials, 2000 pulses, stimulating the left and right ACC respectively.
  Arms: CBT+pseudo-stimulation group
Other: Basic treatment — According to national and international guidelines for the treatment of eating disorders, the basic treatment for patients is nutritional therapy, that is, regular and quantitative dietary treatment, with three regular meals followed by a snack meal 2 hours after the regular meal. Both groups received the same nutritional treatment.

SUMMARY:
The goal of this clinical trial is to learn if dTMS targeting the ACC can be used to rapidly and effectively treat AN. A randomized controlled study design is adopted, in which patients with AN are divided into the CBT+dTMS treatment group and CBT+pseudostimulation group by 1:1 randomization, followed by a 6-week intervention and a half-year follow-up to clarify whether CBT combined with dTMS is superior to single CBT treatment for AN.

DETAILED DESCRIPTION:
The investigators propose hypothesis that CBT improves AN symptoms by modulating the "AN-ACC pathology network", and that high-frequency stimulation targeting the ACC by dTMS can synergize "AN-ACC pathology network" and enhance the efficacy of CBT. In order to verify this hypothesis, a randomized controlled study design is adopted, in which patients with AN are divided into the CBT+dTMS treatment group and CBT+pseudostimulation group by 1:1 randomization, followed by 6-week intervention and a half-year follow up, to clarify the near-term and long-term efficacy and safety of the dTMS treatment. Patients in both groups undergo fMRI examinations, complete delay discounting task (DDT) and body image task before and after each treatment session. Symptoms, psychometrics and side effect questionnaires are followed up at baseline, week 6 (at the end of treatment), and weeks 4, 8, 12 and 24 (after completion of treatment). This study will provide a theoretical and practical basis for the innovative combined intervention method in patients with AN, and to verify the "AN-ACC pathological network" pathomechanism of AN at multiple levels.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Female, aged 18-35 years, right handedness.
* Above primary education.
* Meet the diagnostic criteria of AN in DSM-V, and13.0 kg/m2 ≤ body mass index (BMI)<18.5 kg/m2.
* No systemic nutritional therapy, psychiatric medication or any form of psychotherapy have been received within 1 month before enrollment.
* Able to understand the nature of this study and sign an informed consent form.

Exclusion Criteria:

* Diagnosed with a DSM-5 disease other than anorexia nervosa, or at high risk of suicide, strong impulsive behavior as well as anti-social behavior.
* With severe physical or cognitive impairment.
* Not able to undergo MRI.
* Considered unsuitable for enrollment in this clinical trial for other reasons.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | week 0（baseline）, week 2、week4（during intervention）, week 6（post-intervention）, week10、18、30（follow-up）
  Calculation: BMI = weight (kg) divided by the square of height (m)

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q6.0) | week 0（baseline）, week 2、week4（during intervention）, week 6（post-intervention）, week10、18、30（follow-up）
  Eating Disorder Examination Questionnaire can assess the core symptoms of eating disorders, including behavioral and psychological characteristics, and rate their frequency and intensity, which can assess the severity of the eating disorder. It consists of 4 subscales, including dietary restriction, eating concerns, body image concerns, and weight concerns.
Eating Disorder Inventory (EDI-II) | week 0（baseline）, week 2、week4（during intervention）, week 6（post-intervention）, week10、18、30（follow-up）
  It is a commonly used scale for assessing cognitive-behavioral symptoms of eating disorders and is used to assess the severity of eating disorders. The scale contains 91 items divided into 8 subscales and 3 temporary subscales, including the pursuit of thinness, bulimia, body dissatisfaction, feelings of ineffectiveness, perfectionism, mistrust of others, introspection, maturity fears, abstinence, impulsive regulation and social insecurity.
Beck Depression Inventory (BDI) | week 0（baseline）, week 2、week4（during intervention）, week 6（post-intervention）, week10、18、30（follow-up）
  The BDI consists of 21 items and assesses the patient's accompanying feelings of depression over the past 2 weeks.
Beck Anxiety Inventory (BAI) | week 0（baseline）, week 2、week4（during intervention）, week 6（post-intervention）, week10、18、30（follow-up）
  The Beck Anxiety Inventory (BAI) is a self-rating scale used to assess a patient's anxiety symptoms. The scale consists of 21 items, each evaluating the degree of distress caused by anxiety symptoms. It uses a four-point scale from 1 to 4, with 1 indicating no symptoms and 4 indicating severe symptoms. The total score ranges from a minimum of 21 to a maximum of 84, with higher scores indicating more severe anxiety symptoms.
Self-assessed Compulsive Questionnaire for Eating Disorders (SR-YBC-EDS) | week 0（baseline）, week 2、week4（during intervention）, week 6（post-intervention）, week10、18、30（follow-up）
  The SR-YBC-EDS was developed based on the Yale-Brown Compulsive Questionnaire for Eating Disorders (YBC-EDS), consisting of two parts: the first part is a list of 65 symptomatic items, which is used to identify the subjects' obsessive-compulsive symptoms, and the second part is a list of 8 core items, which is used to assess the frequency and severity of obsessive-compulsive symptoms. All parts contain two dimensions: preoccupation and ritual behavior.
Body Image Tasks | week 0（baseline）, ,week 6（post-intervention）
  Tasks that address excessive concerns about body shape/weight include the following two parts: Body size estimation: The screen will present the above 30 body size pictures sequentially, the subjects will view the body size pictures in 4000ms, and then evaluate the body size of the body pictures in 4000ms, with a score of 1 representing "very low body weight", 4 representing "very overweight", and 4 representing "very overweight". A score of 1 represents "very low weight" and a score of 4 represents "very overweight". Body compare task: The screen will present the above 30 body images in turn, the subjects will have 4000ms to view their own images (with randomized distortions), and then they will have 4000ms to compare their actual body shape with the body shape in the images and assess their emotional level. 1 point represents "very calm" and 4 for "very anxious".
Delay Discounting Task (DDT task) | week 0（baseline）, week 6（post-intervention）
  The study uses a DDT task in a food choice scenario to assess inhibitory impulses. The task requires subjects to make a decision between choosing a small reward in the present or a large reward in the future. Inhibition to choose a small reward in the present implies a strong intertemporal decision-making ability. The task begins with an assessment of their hunger, willingness to eat, and emotional feelings at the moment. Then they are asked to rate 40 pictures of food on a scale of 0 to 10 on five dimensions: familiarity, craving, positive and negative emotions, emotional intensity, and eating control. Pictures of foods with craving scores >7 and eating control <5, as well as matched in familiarity and emotion for use in the ensuing delay discounting task. The choice is made by pressing a button: Patients choosing to get less food immediately are given fewer coupons after the delay. But those waiting for a period of time to get more food are given more coupons after the delay.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Chen, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No